CLINICAL TRIAL: NCT06060509
Title: Effects of Phytosterol-rich Wheat Corn Germ Blended Oil on Immune Function, Oxidative Stress, Serum Metabolites and Intestinal Flora in Dyslipidaemic Population: A Randomised Controlled Trial
Brief Title: Study on the Effects of Wheat and Corn Germ Blend Oil on Antioxidation and Immune Regulation of Dyslipidemia Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Collaborators: Chinese Nutrition Society (Unknown); Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jia-yue Xia, Principal Investigator, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022ZDSYLL031-P02; CNS-NNSRG2021-39 (Other Grant/Funding Number: Chinese Society of Nutrition)
Record Dates: First submitted 2023-09-19; First posted 2023-09-29 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Diseases; Immune System Disorder; Dyslipidemias; Fatty Acid Metabolism Disorder; Oxidative Stress
Keywords: germ blend oil; Gut Microbiota; lipidomics; anti-oxidation; immune regulation; phytosterol
MeSH Terms: conditions — Metabolic Diseases; Immune System Diseases; Dyslipidemias | interventions — Peanut Oil

STUDY DESIGN:
Intervention Model Description: This is a randomised controlled intervention trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The packaging of intervention oil and control oil was consistent, and the subjects could not distinguish what was blend oil and what was control oil. Blinding was also used for outcome assessors, who did not distinguish between the intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wheat corn germ blended oil group (Experimental): Participants in the intervention group replaced the daily cooking oil with wheat and corn germ oil, and were given 25-30 g of cooking oil per day according to the recommended intake of the Chinese Nutrition Society. Lunch and dinner were cooked using a uniform recipe for both intervention and control groups, and breakfast was self-cooked under the uniform dietary guidelines.
  Interventions: Dietary Supplement: Phytosterol-rich Wheat and Corn Germ Blended Oil
- Peanut oil group (Other): Participants in the Peanut oil group replaced the daily cooking oil with Peanut oil, and were given 25-30 g of cooking oil per day according to the recommended intake of the Chinese Nutrition Society. Lunch and dinner were cooked using a uniform recipe for both intervention and control groups, and breakfast was self-cooked under the uniform dietary guidelines.
  Interventions: Dietary Supplement: Peanut oil

INTERVENTIONS:
Dietary Supplement: Phytosterol-rich Wheat and Corn Germ Blended Oil — Blending of corn germ oil and wheat germ oil supplied by Yihai Kerry to obtain germ blended oil with high phytosterol content.
  Arms: Wheat corn germ blended oil group
Dietary Supplement: Peanut oil — Participants in the control group consumed peanut oil daily for cooking.
  Arms: Peanut oil group

SUMMARY:
The goal of this clinical trial is to explore the role of wheat and corn germ blended oils in regulating oxidative stress and immunomodulation in dyslipidaemic populations, to explore their effects on intestinal flora, antioxidant and immunomodulation. The main questions it aims to answer are:

* How does phytosterol-rich wheat corn germ blended oil affect oxidative stress and immune function in dyslipidaemic people compared to peanut oil?
* How does phytosterol-rich wheat corn germ blended oil affect serum metabolites, serum fatty acid profile, and intestinal flora in dyslipidaemic populations compared to peanut oil? What are the specific mechanisms involved?

Participants will be randomly assigned to the intervention and control groups, the packaging of germ oil and peanut oil will have a uniform appearance, and participants will be instructed to replace their household cooking oils with the distributed cooking oil for three months, in addition to replacing all the canteens in the staff units with the trial oil for more than three months. Participants did not know who was the control oil, germ oil or peanut oil, and both were randomly distributed to different groups of participants by the third-party supervisors.

Researchers will compare peanut oil to see if phytosterol-rich germ oil can improve oxidative stress and immune function in dyslipidaemic populations, in addition to exploring possible underlying mechanisms of improvement using multi-omics techniques.

DETAILED DESCRIPTION:
The design of this intervention trial was a randomised controlled trial, in which the included dyslipidaemic population was randomly divided into a wheat corn germ blended oil intervention group and a peanut oil control group, with the male/female ratio, age, and level of basic clinical characteristics balanced between the two groups. The entire test phase consisted of a 14-day washout period and a 3-month intervention period. Participants in the intervention and control groups first entered a 14-day peanut oil washout period, which was followed by a three-month intervention phase. During the intervention phase, two different cooking oils (25-30 g of cooking oil per day according to the recommended intake of the Chinese Nutrition Society) were allocated to the two groups, with peanut oil being consumed by participants in the control group, and germ oil being used to replace the daily cooking oil for participants in the intervention group. After the participants were randomised into groups, they were provided with lunch and dinner according to the Chinese Dietary Guidelines for Residents of China and the local dietary habits of Nanjing, China, and breakfast was provided by the subjects themselves (dietary guidance was given to the subjects during the course of the study, and breakfast recipes were provided uniformly in order to achieve consistency between the two groups), and the intervention period was 3 months. Throughout the project period, all subjects followed their normal dietary habits and maintained a normal level of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65 with BMI less than 30;
* At least one item meets the diagnostic criteria for dyslipidemia (2016 Chinese adult dyslipidemia prevention and treatment guide)
* No serious complications related to liver, kidney, digestive tract, endocrine diseases and chronic diseases;
* Within 3 months, he did not use the drugs and dietary supplements related to reducing blood fat and weight, and agreed not to use the above foods or drugs during the experiment;
* Volunteer to participate in this study after listening to the project introduction and sign the informed consent form.

Exclusion Criteria:

* Pregnant, pregnant or lactating women;
* Patients with liver and kidney dysfunction, diabetes, coronary heart disease, hyperthyroidism, malignant tumor, asthma and other chronic diseases other than dyslipidemia;
* Endocrine disease patients, postoperative patients, patients receiving hormone therapy and psychotic patients;
* Have special eating habits: vegetarian, ketogenic diet (high fat, low carbon water), etc;
* Those who cannot follow the test requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Height in metres | 12 weeks
  Height in metres, physiological parameter
Weight in kilogram | 12 weeks
  physiological parameter
body mass index (BMI) | 12 weeks
  BMI= Weight (kg)/height^2(m)
waist circumference | 12 weeks
  Unit in centimetres,physiological parameter
hip measurement | 12 weeks
  Unit in centimetres,physiological parameter
Systolic blood pressure | 12 weeks
  Units in mmHg. physiological parameter.
diastolic blood pressure | 12 weeks
  Units in mmHg. physiological parameter.
Serum triglyceride concentrations | 12 weeks
  physiological parameter
Serum triglycerides concentrations | 12 weeks
  physiological parameter
Serum LDL cholesterol concentrations | 12 weeks
  physiological parameter
Serum HDL cholesterol concentrations | 12 weeks
  physiological parameter
Percentage of CD3+ total T cells | 12 weeks
  physiological parameter
Percentage of CD4+ T cells | 12 weeks
  physiological parameter
Percentage of CD8+ T cells | 12 weeks
  physiological parameter
Percentage of CD4+ CD8+ cells | 12 weeks
  physiological parameter
Percentage of CD19+ B cells | 12 weeks
  physiological parameter
Percentage of CD16/56+ NK cells | 12 weeks
  physiological parameter
Immunoglobulin G | 12 weeks
  physiological parameter
Immunoglobulin A | 12 weeks
  physiological parameter
Immunoglobulin M | 12 weeks
  physiological parameter
Complement C3 | 12 weeks
  physiological parameter
Immunoglobulin E | 12 weeks
  physiological parameter
reactive oxygen species | 12 weeks
  physiological parameter
superoxide dismutase | 12 weeks
  physiological parameter
malondialdehyde | 12 weeks
  physiological parameter
glutathione | 12 weeks
  physiological parameter

SECONDARY OUTCOMES:
Lipoprotein a | 12 weeks
  physiological parameter
leptin | 12 weeks
  physiological parameter
Transforming growth factor-β | 12 weeks
  physiological parameter
diamine oxidase | 12 weeks
  physiological parameter
endotoxin | 12 weeks
  physiological parameter
Number of participants who smoke | 12 weeks
  questionnaire
Number of participants taking lipid-lowering drugs | 12 weeks
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gui-ju Sun, phD, Study Director — Chinese Nutrition Society
Locations (1):
- Southeast university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There's no plan for that yet.